CLINICAL TRIAL: NCT02331030
Title: A Randomised Controlled Trial Comparing Ultrasound-guided Supraclavicular Brachial Plexus Block With Combined Supraclavicular and Pecs II Block in Patients Undergoing Arteriovenous Grafting Surgery
Brief Title: A Randomised Trial Comparing Supraclavicular Block vs Supraclavicular and Pecs II Block in Arteriovenous Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Kelvin Quek How Yow, Consultant, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014/2047
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Arteriovenous Fistula; Arteriovenous Graft; Kidney Failure, Chronic; Renal Failure, End-stage
Keywords: brachio-axillary; brachio-basilic; interfascial plane block; Pecs II block; supraclavicular brachial plexus block
MeSH Terms: conditions — Arteriovenous Fistula; Kidney Failure, Chronic | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined (C) (Experimental): Ultrasound-guided supraclavicular brachial plexus block with Ropivacaine 0.5% 20ml and Pecs II block with Ropivacaine 0.5% 10ml.
  Interventions: Procedure: Supraclavicular; Procedure: Pecs II block; Drug: Ropivacaine 0.5% 20ml; Drug: Ropivacaine 0.5% 10ml
- Supraclavicular (S) (Active Comparator): Ultrasound-guided supraclavicular BPB with Ropivacaine 0.5% 20ml and sham block (grade 1)
  Interventions: Procedure: Supraclavicular; Procedure: Sham block (Grade 1); Drug: Ropivacaine 0.5% 20ml

INTERVENTIONS:
Procedure: Supraclavicular — Ultrasound-guided supraclavicular brachial plexus block
Procedure: Pecs II block — Ultrasound guided interfascial plane block between pectoralis minor and serratus anterior
  Arms: Combined (C)
Procedure: Sham block (Grade 1) — Sham block -- with skin preparation, ultrasound scanning of pecs II block area, but no actual needle injection
  Arms: Supraclavicular (S)
Drug: Ropivacaine 0.5% 20ml — Local anaesthetic solution administered for supraclavicular block
  Other Names: Naropin
Drug: Ropivacaine 0.5% 10ml — Local anaesthetic solution administered for pecs II block
  Other Names: Naropin
  Arms: Combined (C)

SUMMARY:
This study evaluates the addition of Pecs II block to ultrasound-guided supraclavicular brachial plexus block in patients undergoing arteriovenous graft creation surgery. Participants will be randomised into two equal groups, one receiving supraclavicular and pecs II blocks, the other receiving supraclavicular block and sham block (Grade 1).

DETAILED DESCRIPTION:
Regional anaesthesia (RA) for arteriovenous grafting surgery has advantages of avoiding risks of general anaesthesia (GA) in this group of patients with significant co-morbidities, and beneficial vasodilatation, which may prevent early fistula thrombosis. Hence, RA is preferable to GA for this surgery.

Brachial plexus blocks (BPB) are the most commonly employed RA technique to anaesthetise the upper limb for this surgery. According to the results of a recent 2-year retrospective audit in our centre, ultrasound-guided supraclavicular BPB are the most popular RA technique for this surgery. Anatomically, the T1 and T2 dermatomes are often missed by the supraclavicular BPB. This means that the upper medial arm and axilla (sites involved in brachiobasilic and brachioaxillary arteriovenous grafting) may not be adequately anaesthetised, mandating intraoperative local anaesthetic supplementation by the surgeon. This may affect patients' and surgeons' acceptance of, and satisfaction with the RA technique. The ultrasound-guided Pecs II block, described by Blanco et al, seems to address this problem, as the intercostal T1-6, intercostobrachialis, long thoracic nerves and nerve to serratus anterior are targeted by this block.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for arteriovenous grafting under regional anaesthesia in Changi General Hospital
* American Society of Anaesthesiologists (ASA) physical status 3 to 4
* Elective or emergency surgery

Exclusion Criteria:

* Patients unable to give consent, unable to communicate or cooperate with simple instructions
* Patients with regular consumption of strong opioids (eg. morphine, oxycodone) or steroids
* Patients with allergy or contraindications to local anaesthetics or any of the drugs included in this study
* Patients with pre-existing upper limb neurological deficits
* Patients who refuse or are unsuitable for regional anaesthesia (eg. severely coagulopathic)

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Need for intraoperative local anaesthetic supplementation by the surgeon | Intraoperative
  Whether there was a need for the surgeon to infiltrate a standardised local anaesthetic drug (0.5% ropivacaine) to the operative site during surgery

SECONDARY OUTCOMES:
Volume of intraoperative local anaesthetic supplementation administered | Intraoperative
  Total volume of local anaesthetic drug (0.5% ropivacaine) given by the surgeon
Need for additional sedation or systemic analgesia | Intraoperative
  Whether there was a need for additional sedation or systemic analgesia (on top of what is specified in the protocol)
Highest pain score at Post-Anaesthesia Care Unit (PACU) | Up to 1 hour post-operatively
  Highest pain score on visual analogue scale at the post-anaesthesia care unit
Time to first post-operative analgesia | Up to 24 hours post-operatively
  Duration of time from administration of the block(s) to when patient first requests for oral analgesia. Participants will be followed up for 24 hours after surgery.
Pain score at 12h | 12 hours post-operatively
  Pain score on visual analogue scale 12 hours after surgery
Pain score at 24h | 24 hours post-operatively
  Pain score on visual analogue scale 24 hours after surgery
Patient satisfaction at 24hours | 24 hours post-operatively
  Patient satisfaction with the anaesthesia technique on a 5-point Likert scale 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Quek, MMED (Anaes), Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Confidentiality of individual subjects will be maintained strictly

REFERENCES:
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Arab SA, Alharbi MK, Nada EM, Alrefai DA, Mowafi HA. Ultrasound-guided supraclavicular brachial plexus block: single versus triple injection technique for upper limb arteriovenous access surgery. Anesth Analg. 2014 May;118(5):1120-5. doi: 10.1213/ANE.0000000000000155. PMID 24686046
- [Background] Reynolds TS, Kim KM, Dukkipati R, Nguyen TH, Julka I, Kakazu C, Tokhner V, Chauvapun JP. Pre-operative regional block anesthesia enhances operative strategy for arteriovenous fistula creation. J Vasc Access. 2011 Oct-Dec;12(4):336-40. doi: 10.5301/JVA.2011.8827. PMID 22116664
- [Background] Sahin L, Gul R, Mizrak A, Deniz H, Sahin M, Koruk S, Cesur M, Goksu S. Ultrasound-guided infraclavicular brachial plexus block enhances postoperative blood flow in arteriovenous fistulas. J Vasc Surg. 2011 Sep;54(3):749-53. doi: 10.1016/j.jvs.2010.12.045. Epub 2011 Mar 2. PMID 21367563
- [Background] Purcell N, Wu D. Novel use of the PECS II block for upper limb fistula surgery. Anaesthesia. 2014 Nov;69(11):1294. doi: 10.1111/anae.12876. No abstract available. PMID 25302976
- [Background] Sariguney D, Mahli A, Coskun D. The extent of blockade following axillary and infraclavicular approaches of brachial plexus block in uremic patients. J Clin Med Res. 2012 Feb;4(1):26-32. doi: 10.4021/jocmr723w. Epub 2012 Jan 17. PMID 22383924